CLINICAL TRIAL: NCT04978675
Title: A Prospective Pilot Study Investigating rhPSMA 7.3 PET/MRI in Detecting Recurrent Disease and Aid in Radiotherapy Planning in Patients With Biochemically Recurrent Prostate Cancer
Brief Title: An Investigational Scan (rh PSMA 7.3 PET/MRI) for the Detection of Recurrent Disease and Aid in Radiotherapy Planning in Biochemically Recurrent Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-1347; NCI-2021-05725 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1347 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-07

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Localized Prostate Carcinoma; Prostate Adenocarcinoma
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (F-18 rhPSMA-7.3, PET/MRI) (Experimental): Patients receive F-18 rhPSMA-7.3 IV and after approximately 60 minutes of uptake time, will undergo PET/MRI over 60 minutes. Patients with evidence of F-18 rhPSMA-7.3 disease in the first PET/MRI scan undergo a second F-18 rhPSMA-7.3 PET/MRI at 6 months after the second dose of standard hormonal therapy.
  Interventions: Drug: Fluorine F 18 rhPSMA-7.3; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Fluorine F 18 rhPSMA-7.3 — Given IV
  Other Names: (18F)-rhPSMA-7.3; 18F-rhPSMA-7.3; 18FrhPSMA-7.3; F-18-rhPSMA-7.3; Fluorine F 18 radiohybrid PSMA-7.3; Fluorine-18 rhPSMA-7.3; rhPSMA-7.3 (18F)
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This prospective pilot study will assess the feasibility of rh PSMA 7.3 positron emission tomography/magnetic resonance imaging (PET/MRI) scans in detecting prostate cancer that may have come back (recurrent) in patients with increasing levels of prostate-specific antigen (PSA) following prostate surgery (biochemically recurrent). An increase in PSA levels alone does not tell the doctor where the cancer may be or how much cancer there may be. Imaging tests, like a bone scan, MRI, and/or computed tomography, are often performed to help the doctor learn where or how much cancer there is, and how best to treat the cancer. rhPSMA-7.3 is a radioactive tracer agent that when used with PET/MRI imaging may help diagnose and look for the spread of prostate cancer. Prostate-specific membrane antigen (PSMA) is a protein that is expressed in prostate cancer and this agent targets the PSMA molecule. Giving rh PSMA 7.3 during PET/MRI may help doctors better find where the cancer may be spreading and how much of it there is. The results of this trial may also guide in radiotherapy planning.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the positive predictive value and detection rate of fluorine F 18 rhPSMA-7.3 (F-18 rhPSMA-7.3) positron emission tomography (PET)/magnetic resonance imaging (MRI) in detecting recurrent disease in prostate cancer patients with biochemical recurrence.

SECONDARY OBJECTIVE:

I. To determine the change in salvage radiation treatment plan after F-18 rhPSMA-7.3 PET/MRI imaging.

EXPLORATORY OBJECTIVES:

I. To assess the feasibility of utilizing the PSMA avid recurrent disease on PET/MRI as an alignment tool for MR guided radiotherapy (MR linear accelerator [MR-LINAC]).

II. To assess the treatment response in those patients who demonstrate rhPSMA-7.3 avid disease on the first PET/MRI scan.

OUTLINE:

Patients receive F-18 rhPSMA-7.3 intravenously (IV) and after approximately 60 minutes of uptake time, will undergo PET/MRI over 60 minutes. Patients with evidence of F-18 rhPSMA-7.3 disease in the first PET/MRI scan undergo a second F-18 rhPSMA-7.3 PET/MRI at 6 months after the second dose of standard hormonal therapy.

After completion of study treatment, patients are followed up within 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male and aged > 18 years old
* History of localized adenocarcinoma of the prostate status post (s/p) radical prostatectomy
* An initial elevated PSA >= 0.2 followed by a subsequent confirmatory PSA >= 0.2 clinically suspicious for biochemically recurrent disease
* If the patients were previously taking androgen deprivation therapy (ADT), it should be discontinued at least 12 weeks prior to the study
* Treatment plan includes salvage radiation with or without hormones.
* Patient willing to provide signed informed consent and willing to comply with all required study schedule events, where safe and feasible
* Non-English speaking patients may be enrolled.

Exclusion Criteria:

* Patients with any medical condition or circumstance that the investigator believes may compromise the data collected or lead to a failure to fulfil the study requirements
* Patients who are planned to have an Iodinated contrast agent with computed tomography (CT) or gadolinium based contrast agent with MRI or other PET radiotracer < 24 hours prior to the PET scan
* Patients with contraindication to undergo MRI
* Patients with extreme claustrophobia
* Patients with prior allergy to MRI contrast agent
* Patients who are cognitively impaired

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Positive predictive value (PPV) of F-18 rhPSMA-7.3 positron emission tomography/magnetic resonance imaging (PET/MRI) in detecting recurrent disease | Up to 6 months
  Will be evaluated on both a per-patient and per-region basis. Will estimate the PPV rate and corresponding 95% confidence interval.

SECONDARY OUTCOMES:
Detection rate | Up to 6 months
  Defined as the proportion of patients with prostate-specific membrane antigen (PSMA) positive results. The association between detection and prostate specific antigen level will be assessed by Wilcoxon rank-sum tests.
Change in salvage radiation treatment plan | Baseline up to 6 months
  The proportion of patients with major and minor changes will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Devaki Shilpa S Surasi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT04978675/ICF_000.pdf